CLINICAL TRIAL: NCT03211767
Title: Double-Blind, Randomized, Cross-Over Trial of Aged Garlic Extract for Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Wakunga of America Co. Ltd. (Unknown); Purity Life Health Products LP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HS19581 (B2016:019)
Record Dates: First submitted 2017-01-03; First posted 2017-07-07 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aged garlic extract (Active Comparator): 2 capsules per day containing aged garlic extract
  Interventions: Dietary Supplement: Aged garlic extract
- Placebo (Placebo Comparator): 2 capsules per day without aged garlic extract
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aged garlic extract — Each capsule contains 600mg of aged garlic extract powder
  Arms: Aged garlic extract
Dietary Supplement: Placebo — Each capsule contains cellulose as a filler.
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assess the effect of consumption of aged garlic extract powder on 24 h systolic and diastolic ambulatory blood pressure in hypertensive individuals following 8 weeks of supplementation.

Additional secondary objectives are to assess the effects of aged garlic extract powder intake for 8 weeks on lipid profile (TC, HDL-C, LDL-C, and TG concentrations), blood glucose, office blood pressure, pulse-wave velocity and augmentation index, body mass index, and waist and hip circumference.

DETAILED DESCRIPTION:
Forty hypertensive volunteers between 18 and 75 years will be recruited from the Winnipeg (Manitoba, Canada) area to participate in a two arm crossover, double-blind, randomized, placebo-controlled intervention study for 8 weeks per study period following obtainment of informed consent.

The 2 periods of treatment will include:

1. Treatment period: One capsule twice a day, providing 600 mg each of aged garlic extract powder, for a total of 1200 mg/day of aged garlic extract powder.
2. Control period: The control product will be an identical-looking placebo capsules containing cellulose, which is being used as a filler in the treatment capsules.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent.
* Age: greater than or equal to 40 and less than or equal to 70 years.
* Systolic blood pressure140-160mmHg and/or diastolic blood pressure 90-100 mmHg
* LDL-C less than or equal to 4.9mmol/L
* Those on a stable dose of blood pressure lowering or lipid-lowering medication for greater than or equal to 3 months; if a participant chooses to stop taking blood pressure lowering medications, they will be required to have a minimum 3 month washout period prior to commencement of the study; all other medications medications will be permitted if they are on a stable dose before the start of the study
* Gender: Male and women who are not pregnant (determined by a negative urine pregnancy test at screening for women of childbearing potential) or lactating.
* Language: Participants must be able to read, write and speak English.

Exclusion Criteria:

* Systolic blood pressure > 160mmHg and/or diastolic blood pressure >100mmHg
* Those currently taking (or have taken within the last 3 months) lipid-lowering or blood pressure-lowering supplements (i.e., omega-3 supplements, plant sterols/stanols foods and/or supplements, fibre, etc.)
* Patients with unstable or serious illness, for example, dementia, terminal illness, recent bereavement, secondary hypertension, recent significant medical diagnosis.
* History of cancer, chronic illness, cardiovascular problems, liver and kidney disease (including chronic kidney disease (GFR < 60ml/min/1.732)), diabetes, inflammatory bowel disease, pancreatitis, gallbladder or biliary disease, neurological/psychological disease, bleeding disorders, experienced platelet abnormalities, macrovascular target organ damage (including cerebrovascular disease, stroke, hypertensive retinopathy, left ventricular dysfunction, angina pectoris, myocardial infarction, and peripheral artery disease)
* History of taking any type of garlic preparation (i.e., dried garlic homogenate, aged garlic extract, processed garlic capsule, time-released garlic powder tablet, regular garlic pill, garlic powder and garlic oil) in the past 6 months. in the past 3 months. (Note: regular garlic clove consumption as part of prepared meals, cooking preparations, etc. are permitted throughout the study period)
* Plan to consume any type of garlic preparation (i.e., dried garlic homogenate, aged garlic extract, processed garlic capsule, time-released garlic powder tablet, regular garlic pill, garlic powder and garlic oil. at any time during the study. (Note: regular garlic clove consumption as part of prepared meals, cooking preparations, etc. are permitted throughout the study period)
* Have gained or lost greater than or equal to 10lbs in the previous 3 months, or plan to lose weight at any time during the study
* Plan to become pregnant during the study period.
* Women of childbearing potential not using effective contraception which include: Hormonal contraceptives including combined oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormonal implants; Intrauterine devices (IUD) or Intrauterine system (IUS); Tubal ligation; Vasectomy of partner; Double barrier method (use of physical barrier by both partners, e.g. male condom and diaphragm, male condom and cervical cap)
* Consumption of more than 2 alcoholic drinks/day, or > 14 alcoholic beverages a week, or history of alcoholism or drug dependence.
* History of allergy to garlic, microcrystalline cellulose, silicon dioxide, magnesium stearate, gelatin, hydroxypropylcellulose, or caramel coloring
* Any planned surgeries any time during the study
* Taking medications with psychotropic properties for less than 3 months, i.e., those taking medications with psychotropic properties, such as anti-depressants, anti-anxiety, etc., at a stable consistent dose for a minimum of 3 months are eligible for the study, as long as the medication is consumed at a stable, consistent dose throughout the study period
* Smokers
* Exercising > 15 miles/wk or 4,000 kcal/wk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
24 hour ambulatory blood pressure | 8 weeks

SECONDARY OUTCOMES:
Blood total cholesterol | 8 weeks
Blood low-density lipoprotein cholesterol | 8 weeks
Blood high-density lipoprotein cholesterol | 8 weeks
Blood triglycerides | 8 weeks
Office blood pressure | 8 weeks
Pulse wave velocity | 8 weeks
  Measured by Mobil-O-Graph
Augmentation index | 8 weeks
  Measured by Mobil-O-Graph
Body mass index | 8 weeks
Waist circumference | 8 weeks
Hip circumference | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada